CLINICAL TRIAL: NCT05885048
Title: FertiTOX - Platform for Fertility Related Gonadotoxicity of Cancer Therapies
Brief Title: Impact of Gonadotoxic Therapies on Fertility
Acronym: FertiTOX
Status: Recruiting | Type: Observational
Sponsor: Michael von Wolff (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Michael von Wolff, Prof. Dr. med. Michael von Wolff, Universitätsklinik fur Frauenheilkunde, Inselspital Bern
Organization: Universitätsklinik fur Frauenheilkunde, Inselspital Bern (Other)
Other Study IDs: KEK Bern 2022-02284; KLS 5650-08-2022 (Other: Krebsliga)
Record Dates: First submitted 2023-04-16; First posted 2023-06-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Fertility Issues; Fertility Preservation; Toxicity Due to Chemotherapy; Toxicity Due to Radiotherapy; Effects of Immunotherapy
Keywords: Gonadotoxicity
MeSH Terms: conditions — Neoplasms; Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer female participants: Fertility status before and after gonadotoxic treatment
  Interventions: Diagnostic Test: Blood samples for analysis; Other: Satisfaction evaluation; Other: Quality of Life questionnaire
- Cancer male participants: Fertility status before and after gonadotoxic treatment
  Interventions: Diagnostic Test: Blood samples for analysis; Diagnostic Test: Sperm samples for analysis; Other: Satisfaction evaluation; Other: Quality of Life questionnaire

INTERVENTIONS:
Diagnostic Test: Blood samples for analysis — Test hormone levels in blood
Diagnostic Test: Sperm samples for analysis — Spermiogram
  Groups: Cancer male participants
Other: Satisfaction evaluation — Participant satisfaction assessment
Other: Quality of Life questionnaire — The World Health Organization Quality of Life Brief 26-item Version (WHOQOL-BREF)

SUMMARY:
The goal of this observational study is to learn how gonadotoxic treatments (chemotherapies, radiotherapies or immunotherapies) affect the fertility status of participants with cancer.

The main questions it aims to answer are:

* in females, if cancer therapies reduce the Anti-Müllerian hormone (AMH) concentration (ovarian reserve);
* in males, if cancer therapies reduce sperm concentration (sperm quality).

DETAILED DESCRIPTION:
This is an international multicenter prospective exploratory study of fertility related data generated mostly routinely in fertility centers in Switzerland belonging to the Swiss network "FertiSAVE" as well as in fertility centers in Germany and Austria belonging to the German-Swiss-Austrian network "FertiPROTEKT" and further international centers who are interested to participate. Both networks include in total around 200 centers.

The data, which are mainly part of the routine clinical care, will be collected by the physicians and added to the REDcap study registry. Patients will be coded by the center to be able to follow them up. Each center will only have access to its own registry data set. Access to the total data set is only permitted for the principal investigator and the specific sub-investigators.

Data collection before the start of gonadotoxic treatment will be performed for 5 years.

Data collection after the end of gonadotoxic treatment will be performed for 10 years (time points: at 12-15 months, at 5 years and at 10 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer or with benign reasons undergoing chemotherapy and/or radiotherapy of the pelvis (females) and the testicles (males) and/or immune therapy;
* Willing to participate;
* Austria: 14-50 years old (adolescents and adults), Germany: 18-50 years old, Switzerland: 14-50 years old (adolescents and adults);
* Serum hormone analysis before gonadotoxic therapy (females) or serum hormone analysis and sperm analysis before gonadotoxic therapy (males).

Exclusion Criteria:

* Missing consent;
* Language barrier.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cancer participants from fertility centers (Switzerland, Germany and Austria)
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Müllerian hormone (AMH) concentration in females | Change from baseline in AMH concentration at 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in females (referring to ovarian reserve).
  Blood will be drawn to measure AMH concentration. Unit of measure: for serum AMH value is picomol per liter (pmol/L).
Anti-Müllerian hormone (AMH) concentration in females | Change in AMH concentration at 5 years after time point 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in females (referring to ovarian reserve).
  Blood will be drawn to measure AMH concentration. Unit of measure: for serum AMH value is picomol per liter (pmol/L).
Anti-Müllerian hormone (AMH) concentration in females | Change in AMH concentration at 10 years after time point 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in females (referring to ovarian reserve).
  Blood will be drawn to measure AMH concentration. Unit of measure: for serum AMH value is picomol per liter (pmol/L).
Sperm concentration in males | Change from baseline in sperm concentration at 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in males (referring to sperm quality).
  Participants provide the laboratory with a sperm sample for analysis. Unit of measure: for sperm concentration is millions per milliliter (10^6/mL).
Sperm concentration in males | Change in sperm concentration at 5 years after time point 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in males (referring to sperm quality).
  Participants provide the laboratory with a sperm sample for analysis. Unit of measure: for sperm concentration is millions per milliliter (10^6/mL).
Sperm concentration in males | Change in sperm concentration at 10 years after time point 12-15 months after the end of gonadotoxic treatment
  Fertility status after gonadotoxic treatment in males (referring to sperm quality).
  Participants provide the laboratory with a sperm sample for analysis. Unit of measure: for sperm concentration is millions per milliliter (10^6/mL).

SECONDARY OUTCOMES:
Fertility preservation measures performed | Before the start of gonadotoxic treatment
  Proportion of female participants who freeze their ovarian tissue, oocytes, zygotes or embryos.
  Proportion of male participants who freeze their sperm or testicular tissue.
Satisfaction with the fertility preservation counselling before the gonadotoxic treatment | 12-15 months after the end of gonadotoxic treatment
  Both female and male participants will have to rate their counselling satisfaction by choosing a score on a scale from 1 to 10. Value 1, being the lowest score (not satisfied at all) and value 10 being the highest score (very satisfied).
Satisfaction with the decision to have undergone fertility preservation measures or not | 12-15 months after the end of gonadotoxic treatment
  Both female and male participants will have to rate their decisional satisfaction by choosing a score on a scale from 1 to 10. Value 1, being the lowest score (not satisfied at all) and value 10 being the highest score (very satisfied).
Number of spontaneous pregnancies and children born | 12-15 months, 5 years and 10 years after the end of gonadotoxic treatment
  Pregnancies which occured naturally, without the help of fertility preservation measures.
Number of pregnancies and children born with the help of fertility preservation measures | 12-15 months, 5 years and 10 years after the end of gonadotoxic treatment
  Pregnancies which occured with the help of fertility preservation measures (in females: frozen ovarian tissue, oocytes, zygotes or embryos, and in males: frozen sperm or testicular tissue).
Quality of life assessment | 12-15 months, 5 years and 10 years after the end of gonadotoxic treatment
  The World Health Organization Quality of Life Brief 26-item version (WHOQOL-BREF) is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items), while the remaining two items are for the overall QoL and general health domains.

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Wolff, Prof. Dr., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Women's Hospital (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Wolff M, Germeyer A, Bottcher B, Magaton IM, Marcu I, Pape J, Sanger N, Nordhoff V, Roumet M, Weidlinger S. Evaluation of the Gonadotoxicity of Cancer Therapies to Improve Counseling of Patients About Fertility and Fertility Preservation Measures: Protocol for a Retrospective Systematic Data Analysis and a Prospective Cohort Study. JMIR Res Protoc. 2024 Mar 20;13:e51145. doi: 10.2196/51145. PMID 38506900
- [Background] Weidlinger S, Graber S, Bratschi I, Pape J, Kollar A, Karrer T, von Wolff M. A Systematic Review of the Gonadotoxicity of Osteosarcoma and Ewing's Sarcoma Chemotherapies in Postpubertal Females and Males. J Adolesc Young Adult Oncol. 2024 Aug;13(4):597-606. doi: 10.1089/jayao.2023.0185. Epub 2024 Apr 17. PMID 38629685
- See also: A platform for gonadotoxicity of cancer therapies — https://fertitox.com/
- Available data/document: Study Protocol — https://www.researchprotocols.org/2024/1/e51145